CLINICAL TRIAL: NCT07347756
Title: The Effect of Gait Imagery on the Muscular Activity of Lower Limbs and Lower Body Kinematics in Subacute Stroke Survivors
Brief Title: The Effect of Gait Imagery on the Muscular Activity of Lower Limbs and Lower Body Kinematics in Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hana Haltmar (Other)
Responsible Party: Sponsor-Investigator, Hana Haltmar, Clinical Researcher, Palacky University
Organization: Palacky University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IGA_FTK_2021_014; 13/2021 (Other: Faculty of Physical Culture Palacky University Olomouc)
Record Dates: First submitted 2025-12-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Motor Imagery; Stroke
Keywords: motor imagery; gait; surface electromyography; angular velocity; acceleration; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All individuals will be instructed to realize normal gait imagery (NGI) and gait on the line imagery (GLI) modalities in a single experimental session. The order of imagining these two gait modalities was randomized and both modalities consisted of these tasks: rest (non-imagery task), NGI/GLI before and after the real execution of normal gait/tandem gait on the line. The order of the tasks was not randomized.
  Individuals are also asked about the ease/difficulty of imagining both NGI/GLI before and after the real execution of gait tasks using a five-point scale.
  Each task is measured once for 30 s with respect to sustained attention and possible onset of fatigue.
  Interventions: Behavioral: gait imagery

INTERVENTIONS:
Behavioral: gait imagery — The initial position, which is identical for all measured tasks, consisted of an upright bipedal stance in front of an unobtrusive white screen with feet at pelvic width, upper limbs held loosely along the body, eyes open and facing forward. During the rest task, non-motor imagery task, participants are instructed to sing the song "Happy Birthday" in their minds.
  NGI before the real execution of normal gait and GLI before the real execution of gait on the line are tasks associated with the imagery of normal gait or tandem gait on the line. Participants first observed a 5 m section of the corridor for NGI, or a line located in the middle of the same corridor for GLI.
  The last tasks, NGI after the real execution of normal gait and GLI after the real execution of gait on the line, differed from above mentioned tasks in the immediate real experience of normal gait or gait on the line.

SUMMARY:
The aim of the study is to evaluate the effect of normal gait imagery and gait on a line imagery on lower limb muscle activity and lower body kinematics in stroke survivors.

DETAILED DESCRIPTION:
Gait imagery is a cognitive process involving the mental simulation of a gait that is not actually performed. According to current studies, gait imagery has very similar neural activity to that observed in real gait. This activity can be observed not only at the central level, but also at the end effector - the muscle - using surface electromyography. Across studies, muscle activity and kinematics are evaluated in particular when imagining analytical movements of the upper or lower limbs, but complex and posturally more demanding movements (in our case, gait and its modification - gait on a line) are studied to a lesser extent. Independent walking and the ability to adapt it to the terrain is important in rehabilitation therapy for patients with limited mobility. These individuals include, among others, a stroke survivors. The aim of the study is therefore to evaluate the effect of normal gait imagery and gait on a line imagery on lower limb muscle activity and lower body kinematics in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subacute stage (1 week - 2 months after the onset of the attack) after primary attack of stroke
* Ischemic origin of stroke
* Good cognitive level to understand the study
* Minimum age of 18 years
* Clinically manifested hemiparetic gait with ability to perform independent walking for at least five minutes
* Mild motor deficit with ability to maintain standing without any support
* Ability to walk independently without any manual assistance of another person (≥ 3/5 points according to the Functional Ambulation Categories)
* Good level (≥ 4/7 points) of kinesthetic and visual MI according to the Czech version of the MIQ-RS questionnaire

Exclusion Criteria:

* Present impairments in communication and cognition
* An additional neurological, internal, psychological or psychiatric disorder or severe musculoskeletal disorder that may affect the ambulation
* Previous experience with MI
* Pain during the measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Objective measurement of muscle activity | Day 1
  Muscle activity [V] will be measured by surface electromyography during all tasks (rest and gait imagery before/after real gait execution) across both gait imagery modalities (normal gait imagery and gait on the line imagery).
Objective measurement of lower body kinematics 1 | Day 1
  Lower body kinematics will be measured by gyroscope [deg/s] during all tasks (rest and gait imagery before/after real gait execution) across both gait imagery modalities (normal gait imagery and gait on the line imagery).
Objective measurement of lower body kinematics 2 | Day 1
  Lower body kinematics will also be measured by accelerometer [g] during all tasks (rest and gait imagery before/after real gait execution) across both gait imagery modalities (normal gait imagery and gait on the line imagery).

SECONDARY OUTCOMES:
Questionnaire - Evaluation of gait imagery | Day 1
  Individuals will be asked about ease/difficulty of imagining both normaI gait imagery/gait on the line imagery before and after the real execution of gait tasks using a five-point scale (maximum value - 5 points [easy] to minimum value - 1 point [difficult]).

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Palacky University, Olomouc
  - University Hospital Olomouc, Olomouc

REFERENCES:
- [Result] Haltmar H., Janura M., Haltmar M., & Elfmark M. (2024).The effect of gait imagery and its more demanding variant on muscle activity in stroke survivors. Rehabilitace a fyzikální lékařství, 31(3), 116-125. doi: 10.48095/ccrhfl2024116.
- See also: This article describe how muscle activity of selected paretic and non-paretic lower limb muscles changes in subacute stroke survivors when imagining normal gait and its more challenging variant, gait on the line. — https://redakce.carecomm.cz/rhfl/cs/article/view/2260/886